CLINICAL TRIAL: NCT03417973
Title: A Prospective Single-arm, Multi-center Clinical Study Examining Quality of Life and Pain Following Dorsal Root Ganglion Stimulation for the Treatment of Chronic Intractable Pelvic and Lower Limb Pain
Brief Title: Quality of Life and Pain Changes Due to DRG Stimulation for Chronic Pain
Acronym: ACTIVE
Status: Terminated | Type: Observational
Why Stopped: Sponsor withdrew funding
Sponsor: KM Clinical Research Group (Industry)
Responsible Party: Principal Investigator, Kate McLellan, Principle Investigator, KM Clinical Research Group
Other Study IDs: 2017-PN-01
Record Dates: First submitted 2017-08-11; First posted 2018-01-31 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Spinal; Nerve Root, Pain; Pelvic Pain; Regional Pain Syndrome; Chronic Pain Syndrome; Complex Regional Pain Syndromes
Keywords: dorsal root ganglion
MeSH Terms: conditions — Pain; Pelvic Pain; Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- complex regional pain syndrome: Chronic regional pain of lower limb(s) patients medically indicated to have dorsal root ganglion (DRG) stimulation for control of pain. DRG stimulator will be implanted for trial of 3-4 days and then permanently, if patient find acceptable levels of pain control with trial.
  Interventions: Device: dorsal root ganglion neuromodulation
- Chronic pelvic pain: Chronic pelvic or urological pain patients medically indicated to have dorsal root ganglion (DRG) stimulation for control of pain. DRG stimulator will be implanted for trial of 3-4 days and then permanently, if patient find acceptable levels of pain control with trial.
  Interventions: Device: dorsal root ganglion neuromodulation

INTERVENTIONS:
Device: dorsal root ganglion neuromodulation — stimulation for neuromodulation of the dorsal root ganglion

SUMMARY:
ACTIVE study- a prospective observational clinical study examining the changes in quality of life and pain following dorsal root ganglion stimulation for the treatment of chronic intractable pelvic and lower limb pain.

DETAILED DESCRIPTION:
Objectives The primary objective is changes in pelvis and/or lower limb pain following dorsal root ganglion (DRG) stimulation. Pain levels will be determined using a 10-point Visual Analog Scale (VAS) with 10= Extreme Pain and 0= No Pain.

The null hypothesis is there will be no change in the subjects' self-reported pain levels from baseline to 52 weeks post-stimulator implantation. The alternate hypothesis is a significant change in pain levels.

Secondary objectives include changes in physical health, quality of life, and pain-related prescription medication usage. Each subject's overall quality of life will be measured with the National Institute of Health's PROMIS Global Health survey v1.2. Physical activity changes will be assessed using the NIH PROMIS Pain Interference 6a SF v1.0 and Pain Intensity 3a scale v1.0. Finally, patients will be asked the name, dosage, and frequency of use of any pelvic and/or lower limb pain-related prescription medications they are currently using.

Design and Outcomes This is a prospective observational single-arm study to access the primary outcome variable of pelvic and/or lower limb pain Intervention and Duration There will be no study intervention. Subjects will only be monitored and evaluated for pre and post-operative pain, physical activity levels, quality of life, and medication use. Subjects will be followed for 12 months following their DRG stimulation implant surgery.

Sample Size and Population This study will last for 4 years starting July 1, 2017. There will be no maximum subject population size. We aim for a minimum population size of 500 in order to give statistical significance with results. Subjects will be stratified by area of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed orthopedic surgery or procedure by their healthcare provider.
* Previous conservative care such as physical therapy or chiropractic care that failed to provide adequate pain relief.
* Willing and able to adhere to the protocol of the study including the survey timeline.
* Between the ages of 18-85 years.

Exclusion Criteria:

* Inability or unwillingness to give written informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients medically indicated to receive DRG stimulator for treatment of chronic lower limb and/or pelvic pain.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in pain | 12 months post-permanent dorsal root ganglion stimulator implantation
  change in visual analogue scale rating

SECONDARY OUTCOMES:
Change in quality of life | 12 months post-permanent dorsal root ganglion stimulator implantation
  change in NIH PROMIS Global health v2 score
Change in physical health | 12 months post-permanent dorsal root ganglion stimulator implantation
  Change in Pain Behavior and Pain Interference measures

OTHER OUTCOMES:
Change in pain-related prescription medication use | 12 months post-permanent dorsal root ganglion stimulator implantation
  change in self-reported medication usage and types of medications needed to control pain

CONTACTS AND LOCATIONS:
Overall Officials: Kate McLellan, PhD, Principal Investigator — KM Clinical Research Group
Locations (1):
- KM Clinical Research Group, Murrieta, California, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers will only see participation data for the subjects they recruit and enroll in the study.